CLINICAL TRIAL: NCT06895681
Title: UCSF Biobank for Studying Hereditary Cancers and Tumor-Associated Mutations
Brief Title: UCSF Biobank for Hereditary Cancers and Tumor-Associated Mutations
Status: Not yet recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 24986
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor; Solid Tumor, Adult; Somatic Mutation; Solid Tumor, Unspecified, Adult; Hereditary Cancer
Keywords: Germline Mutations; Tumor-Associated Mutations
MeSH Terms: interventions — Blood Specimen Collection; Histocompatibility Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Participant-derived tissue, blood, ascites fluid, and pleural fluid samples will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with solid tumor malignancies: Participants' biospecimen samples (Tissue, Excess fluid (i.e., ascites, pleural effusions, and Blood) will be obtained during non-study, routine medical visits whenever possible, to minimize participant risk. Blood samples will be collected up to 5 times from consenting participants.
  Interventions: Procedure: Blood Sample; Procedure: Tissue Sample; Procedure: Excess fluid Sample; Other: Medical Chart Review

INTERVENTIONS:
Procedure: Blood Sample — Obtained at the time of non-study related routine blood draw.
  Other Names: Blood Specimen
Procedure: Tissue Sample — Obtained at the time of non-study related routine biopsy or surgical procedure.
  Other Names: Tissue Specimen
Procedure: Excess fluid Sample — Obtained at the time of non-study related routine biopsy, surgical procedure, paracentesis, or thoracentesis procedure.
Other: Medical Chart Review — Demographic, clinical, and pathologic information will be extracted from the medical record
  Other Names: Medical Record Review

SUMMARY:
This is a non-therapeutic clinical research biorepository protocol designed to obtain, store, and clinically annotate biospecimens from participants with hereditary cancers. Those biospecimens will be used to generate participant-derived tumor models that will serve as a resource to better understand hereditary cancers and develop new efficient therapies.

DETAILED DESCRIPTION:
Primary Objective:

1. To generate a repository of participant-derived tumor models* and specimens** - annotated with demographic, clinical, and pathologic data - from adults with solid tumor malignancies with germline or somatic tumor-associated mutations and/or a personal or family history of cancer.

   * Participant-derived models may include (but are not limited to) xenografts (PDX), organoids (PDO), and cell lines (PDCLs).

     * Specimens may include tissue, ascites and pleural fluid, and blood.

Exploratory Objectives

1. To correlate in vivo drug sensitivity of participant-derived models with patient clinical response.
2. To conduct blood-based assessment of tumor-associated biomarkers (DNA/RNA/protein, etc.).
3. To describe tumor and blood-based biomarkers that are predictive of clinical response.
4. To correlate changes in tumor and blood-based biomarker expression with clinical outcomes over time.
5. To perform genomic and transcriptomic profiling of banked specimens and correlate findings with clinical outcomes, prognostic markers, and biomarkers.
6. Unspecified cancer-centric research in the Munster Lab and other future unspecified research.

OUTLINE:

Participants will have biospecimens collected at non-study, routine procedures or visits to be stored at UCSF. Specimens will be processed and banked as per standard operating procedure. Participants will be followed through medical record chart review for a period of 10 years after signing informed consent, and be contacted every 3 months (± 2 months) for the first year and every 6 months (± 3 months) thereafter to allow updates to health status.

ELIGIBILITY:
Inclusion Criteria:

For participants undergoing collection of tissue, ascites, and/or pleural effusions:

1. Ability to understand and willingness to voluntarily sign a written informed consent document prior to any study-related assessments or procedures are conducted.
2. Individuals 18 years of age or older on the day of signing informed consent.
3. Individuals with solid tumor malignancy with germline or somatic cancer-associated mutations and/or Individuals with a family history or personal history of cancer.
4. Must be planning to undergo one of the following procedures as part of their routine care (or as a research procedure under a UCSF-sponsored IIT protocol):

   1. Surgical resection
   2. Biopsy (open, incisional, excisional, punch, core needle, and/or fine needle aspiration (FNA) are all permitted)
   3. Paracentesis
   4. Thoracentesis

For participants undergoing blood banking:

1. Ability to understand and willingness to voluntarily sign a written informed consent document prior to any study-related assessments or procedures are conducted.
2. Individuals 18 years of age or older on the day of signing informed consent.
3. Individuals with a family history or personal history of cancer.
4. Must be planning to undergo a blood draw as part of their routine care (or as a research procedure under a University of California, San Francisco (UCSF) -sponsored investigator-initiated trial (IIT) protocol); or willing to undergo an additional blood draw outside of their routine care.

Exclusion Criteria:

1. Known history of HIV, Hepatitis B, or Hepatitis C (as documented in the medical record) or other infectious disease that in the judgment of the investigator could pose a risk to research personnel or mice, or negatively impact Patient derived xenografts (PDX) tumor engraftment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with solid tumor malignancies and germline or somatic mutations for cancer and/or a personal or family history of cancer
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Develop participant-derived tumor models of hereditary cancers | Up to 10 years
  Participant-derived models may include (but are not limited to) xenografts (PDX), organoids (PDO), and cell lines (PDCLs). These models recapitulate the biology and tissue context of the original tumors from which they are derived and can be used to study effective therapeutic strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Munster, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No